CLINICAL TRIAL: NCT07118969
Title: A Semi-Experimental Study on Improving University Students' Knowledge and Awareness of Breast Cancer
Brief Title: A Quasi-Experimental Study to Improve Breast Cancer Awareness Among University Students
Acronym: BCAwarenessUni
Status: Active, not recruiting | Type: Observational
Sponsor: Mardin Artuklu University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Kadriye Olgac, Research Assistant, Mardin Artuklu University
Other Study IDs: MAU-HEM-KO-01; 1919B012414986 (Other Grant/Funding Number: TÜBİTAK)
Record Dates: First submitted 2025-08-01; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Awareness; Health Education; Early Detection of Cancer
Keywords: Breast Cancer Awareness; Breast Cancer Knowledge; Breast Self-Examination (BSE); Cancer Screening; Early Detection of Cancer; Health Education; University Students; Preventive Health Behavior
MeSH Terms: conditions — Health Education; Breast Self-Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female Student: Female students aged 18 years and older enrolled at Mardin Artuklu University. A total of 100 participants will be selected through cluster sampling from five faculties (Faculty of Literature, Faculty of Economics and Administrative Sciences, Faculty of Islamic Sciences, Faculty of Tourism, and School of Physical Education and Sports). Participants will receive a five-session breast cancer education program, and their knowledge and awareness levels will be assessed before and two months after the training.
  Interventions: Other: Breast Cancer Awareness Training

INTERVENTIONS:
Other: Breast Cancer Awareness Training — A structured breast cancer education program consisting of five sessions, each lasting 90 minutes. The program covers breast cancer risk factors, early detection methods including breast self-examination (BSE), clinical breast examination, mammography, and health-promoting behaviors. The sessions are conducted in group settings within university faculties. The education aims to increase participants' knowledge and awareness of breast cancer and encourage early detection practices.

SUMMARY:
Breast cancer is one of the most common cancers among women worldwide and a leading cause of cancer-related deaths. Despite advances in early detection and screening methods, breast cancer remains a significant public health issue, especially in populations with low awareness levels.

This study aims to evaluate the effect of a breast cancer education program on the knowledge and awareness of female students at Mardin Artuklu University. The study will include 100 voluntary female students aged 18 and older from five faculties, selected using cluster sampling.

Participants will complete a Personal Information Form, the Comprehensive Breast Cancer Knowledge Test, and the Breast Cancer Awareness Scale before the intervention. They will then attend a five-session breast cancer education program, with each session lasting 90 minutes. A post-test will be administered two months after the completion of the training.

The education program is expected to improve students' knowledge and awareness of breast cancer, encourage early detection behaviors, and contribute to the prevention and early diagnosis of breast cancer.

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignancies among women worldwide and remains a major public health problem and a leading cause of cancer-related deaths. Despite advancements in healthcare systems, screening programs, and early detection methods, breast cancer continues to pose a significant threat, particularly in populations with low awareness levels. Early detection, including breast self-examination (BSE), clinical breast examination, and mammography, is crucial and is strongly associated with individuals' knowledge and awareness.

The literature indicates that young women, particularly university students, often lack sufficient knowledge about breast cancer and have limited awareness regarding early detection and screening behaviors. University students represent a critical target group for health education, as they are at an age where adopting preventive health behaviors and gaining accurate knowledge can have a long-term positive impact. Therefore, implementing educational programs to increase young women's knowledge and awareness of breast cancer is expected to improve early detection rates and contribute to the reduction of breast cancer mortality in the long term.

This study is a quasi-experimental, single-group, pre-test-post-test design to be conducted among female students at Mardin Artuklu University. The study population will include 100 female students enrolled in the 2025-2026 academic year. Cluster sampling will be used, and 20 students will be selected from each of the following faculties: Faculty of Literature, Faculty of Economics and Administrative Sciences, Faculty of Islamic Sciences, Faculty of Tourism, and School of Physical Education and Sports.

Prior to the educational intervention, participants will complete a Personal Information Form, the Comprehensive Breast Cancer Knowledge Test, and the Breast Cancer Awareness Scale. Following this, a five-session breast cancer education and awareness program will be implemented. Each session will last 90 minutes and will cover breast cancer risk factors, early detection methods, steps of BSE, and health-promoting behaviors. Two months after the completion of the educational program, a post-test will be administered to evaluate changes in knowledge and awareness.

This study is expected to enhance university students' knowledge and awareness of breast cancer, encourage regular early detection and screening practices, promote healthy lifestyle behaviors, and contribute to the early diagnosis and prevention of breast cancer in Türkiye. The findings may provide valuable guidance for developing similar educational interventions in the field of public health nursing.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be students at Mardin Artuklu University.

Exclusion Criteria:

* Students with any physical or mental health issues
* Individuals with a diagnosis or history of mental illness will be excluded from the study.

Min Age: 18 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women
Study Population: The research population will consist of 100 students enrolled at Mardin Artuklu University in the 2025-2026 academic year. Female students over the age of 18 who are willing to participate will be included in the study. The study will be conducted using cluster sampling, involving five faculties at Mardin Artuklu University-the Faculty of Literature, the Faculty of Economics and Administrative Sciences, the Faculty of Islamic Sciences, the Faculty of Tourism, and the School of Physical Education and Sports-with 20 students from each faculty.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-02-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Change in Breast Cancer Knowledge | Baseline and 2 months post-intervention
  Change in scores on the Comprehensive Breast Cancer Knowledge Test before the education program and two months.
  As scores increase, breast cancer knowledge and awareness increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Artuklu Unıversity, Mardin, Artuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data contain personally identifiable information and will not be shared to protect participant privacy. The study is limited to a single institution and data will only be used for internal academic purposes. De-identified data will not be shared as this study is for educational purposes only.